CLINICAL TRIAL: NCT05325762
Title: Effect of Propofol on Postoperative Sleep Quality in Elderly Patients With Sleep Disorders: a Multicentre, Randomized, Controlled Clinical Study
Brief Title: Effect of Propofol on Postoperative Sleep Quality in Elderly Patients With Sleep Disorders
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XiangyaH1
Record Dates: First submitted 2022-02-27; First posted 2022-04-13 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-02

CONDITIONS: Sleep Disorder
Keywords: Sleep Disorder; Propofol; Dexmedetomidine
MeSH Terms: conditions — Sleep Wake Disorders | interventions — Propofol; Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Patients were evaluated with MOAA/S by intravenous administration of propofol, dexmedetomidine, or normal saline until successful sleep (MOAA/S≤2)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The blind group included the principal investigator, and any other participants in the recording, evaluation, analysis, or review of efficacy/safety endpoint data, who were primarily responsible for study operations other than drug administration (e.g., subject screening, efficacy and safety indicator recording, statistical analysis, etc.).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Propofol (Experimental)
  Interventions: Drug: Propofol
- Dexmedetomidine (Active Comparator)
  Interventions: Drug: Dexmedetomidine
- saline (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Propofol — At 21:00 on the night of tracheal extubation, propofol was administered intravenously with a microinjection pump for 2min. MOAAS/S was used to evaluate subjects 30 seconds after the end of administration.
  Arms: Propofol
Drug: Dexmedetomidine — Dexmedetomidine was at 21 PM on the day of tracheal extubation: Dexmedetomidine was injected intravenously beginning at 00. During administration, patients were evaluated with MOAA/S every 2min.
  Arms: Dexmedetomidine
Drug: Saline — At 21:00 PM on the day of tracheal extubation, normal saline was injected intravenously. During the administration, patients were evaluated with MOAA/S every 2 minutes.
  Arms: saline

SUMMARY:
This study intends to conduct postoperative sleep intervention for elderly patients with sleep disorders undergoing surgery. We hope to explore whether propofol can improve the postoperative sleep quality of elderly patients with sleep disorders, prevent the occurrence of postoperative delirium in elderly patients, relieve patients' pain, promote patients' postoperative rehabilitation, and provide reference for realizing the rapid rehabilitation of elderly patients with sleep disorders through intravenous administration of research drugs, on the premise of improving patient comfort and ensuring patient safety.

DETAILED DESCRIPTION:
The purpose of this multicenter, randomized, controlled clinical study was to evaluate the efficacy and safety of propofol compared with normal saline and dexmedetomidine in the effect of postoperative sleep quality in elderly subjects with sleep disorders. Subjects were randomly assigned to propofol group, dexmedetomidine group or normal saline control group. Propofol group: At 21:00 on the night of tracheal extubation, propofol was administered intravenously. MOAAS/S was used to evaluate subjects 30 seconds after the end of administration.Dexmedetomidine group: treated with dexmedetomidine at 21 PM on the day of tracheal extubation. During administration, patients were evaluated with MOAA/S every 2min. Normal saline control group: 21 on the night of tracheal extubation: Normal saline was injected intravenously at the rate of 0.5ml/(kg.h) beginning at 00. During the administration, patients were evaluated with MOAA/S every 2min. The effect of drugs on sleep improvement was evaluated by subjective scale and objective electrical monitoring.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 60 years old
* Chronic insomnia
* Pittsburgh Sleep Quality Index>5 points
* Daytime functional impairment (component Ⅶ ≥2 points in PSQI)
* Patients undergoing elective surgery
* Patients to be admitted to ICU after surgery
* Voluntarily participate in the study and sign the informed consent

Exclusion Criteria:

* Subjects with severe hemodynamic instability
* Subjects with difficult airway
* Patients with other sleep disorders (including sleep apnea syndrome, exercise-related sleep disorders and other types of sleep disorders)
* Subjects requiring sedation, mechanical ventilation, or sleep prior to medication;
* Severe liver dysfunction (Child-Pugh GRADE C)
* Severe renal dysfunction (requiring dialysis before surgery)
* Patients with allergies to study drugs and related ingredients
* Patients with severe dementia, low cognitive function, language impairment, severe hearing or vision impairment, mental disorder, coma and other conditions cannot complete the assessment

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-10-25 (Estimated); Study Completion 2023-12-25 (Estimated)

PRIMARY OUTCOMES:
Sleep improvement efficiency | Preoperative, postoperative 1-7 days, postoperative 30 days
  The total score of The Leeds Sleep Evaluation Questionaire was > 100 （The score ranges from 0 to 100， a higher scores mean a better outcome.）, the incubation period of sleep was < 30min, the sleep duration was > 5h, and the sleep quality was good. Assess changes at several points in time.

SECONDARY OUTCOMES:
Safety of drug use | The first night after surgery
  Adverse events and serious adverse events.
Sleep scale assessment | Preoperative, postoperative 1-7 days, postoperative 30 days
  Preoperative and postoperative sleep was assessed using Pittsburgh sleep quality index. Assess changes at several points in time.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - West China Hospital, Sichuan University, Chengdu, Sichuan